CLINICAL TRIAL: NCT03370380
Title: Intravitreal Aflibercept in Patients With Retinal Pigment Epithelial Detachment (PED) Secondary to Age Related Macular Degeneration (AMD)
Brief Title: Aflibercept in Patients With Pigment Epithelial Detachments (PED)
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: AMD-PEA 14
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Pigment Epithelial Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — aflibercept

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aflibercept — Patients are treated according to authorization of Aflibercept

SUMMARY:
Uncontrolled single site non randomized non interventional study to determine the safety and efficacy of intravitreal injections of Aflibercept in patients with recent vision loss due to retinal pigment epithelial detachment secondary to AMD

ELIGIBILITY:
Inclusion Criteria:

* Patients with vascular PED due to AMD
* Male or female patients with the age > 50 years
* Angiographic and via OCT ensured PED ≥ 200 µm in the eye for treatment
* Written informed consent
* Best corrected visual acuity (ETDRS-Visus): 24 - 73 letters within

Exclusion Criteria:

* Patients that do not fulfill the a. m. inclusion criteria
* Patients which have been treated with steroids or with verteporfin via photodynamic therapy or focal lasercoagulation treatment until 3 months before,
* Anti VEGF therapy until 1 month before screening
* Patients with other retinal vascular diseases including diabetic rethinopathia or retinal vein occlusion
* Other ocular operative procedurs 3 months before Screening
* Anamnesis of non controlled glaucoma
* Active or intraocular Inflammation or Inflammation of ocular adnexa
* Subfoveal fibrosis within study eye
* Larger surgical interventions 1 month before Screening
* Anamnesis of serious cardiovascular diseases or stroke 6 months before srceening
* Allergy of components of the study medication
* Patients which might be not compliant
* Patients participating at another clinical trial at the same time
* Pregnancy, breastfeeding, women in child-bearing years without using a safe contraception method
* Chronical alcohol- or drug abuse within the last year
* lack of capacity and/or knowledge of German language
* Neurologic disease i. e. multiple sclerosis

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: In total 20 eyes/patients are treated and observed after inclusion diagnosis and informed consent over a period about 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-04-17 (Actual); Primary Completion 2018-04-23 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Retention and improvement of visual acuity | Screening until 1 month after last injection within study eye (Month 12)
  Visual acuity after treatment completion compared to baseline
Height of Pigment Epithel Detachment | Screening until 1 month after last injection within study eye (Month 12)
  The height of PED after treatment completion compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Clemens, Dr. med., Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Clemens CR, Alten F, Termuhlen J, Mihailovic N, Rosenberger F, Heiduschka P, Eter N. Prospective PED-study of intravitreal aflibercept for refractory vascularized pigment epithelium detachment due to age-related macular degeneration: morphologic characteristics of non-responders in optical coherence tomography. Graefes Arch Clin Exp Ophthalmol. 2020 Jul;258(7):1411-1417. doi: 10.1007/s00417-020-04675-y. Epub 2020 Apr 18. PMID 32306096